CLINICAL TRIAL: NCT00791388
Title: Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of PG 760564 Administered Twice Daily to Healthy Male and Female Volunteers for 14 Days (27 Doses).
Brief Title: Multiple Rising Oral Dose Study of PG 760564 Administered Twice Daily to Healthy Male/Female Volunteers for 14 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: William S Aronstein, PhD, MD, Procter and Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2005046
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- placebo (Placebo Comparator): placebo capsule
  Interventions: Drug: Placebo
- 50 mg PG 760564 (Experimental): 50 mg PG 760564 active
  Interventions: Drug: PG-760564
- 100 mg PG 760564 (Experimental): 100 mg PG 760564 active
  Interventions: Drug: PG-760564
- 200 mg PG 760564 (Experimental): 200 mg PG 760564 active
  Interventions: Drug: PG-760564
- 400 mg PG 760564 (Experimental): 400 mg PG 760564 active
  Interventions: Drug: PG-760564

INTERVENTIONS:
Drug: Placebo — oral capsule, 2x/day for 14 days
  Arms: placebo
Drug: PG-760564 — oral capsule, 50 mg, 2x/day for 14 days
  Arms: 50 mg PG 760564
Drug: PG-760564 — oral capsule, 100mg, 2x/day for 14 days
  Arms: 100 mg PG 760564
Drug: PG-760564 — oral capsule, 200 mg, 2x/day for 14 days
  Arms: 200 mg PG 760564
Drug: PG-760564 — oral capsule, 400 mg, 2x/day for 14 days
  Arms: 400 mg PG 760564

SUMMARY:
This study is a multiple ascending dose study to Assess the Safety, Tolerability, and Pharmacokinetics of orally dosed PG 760564 Administered Twice Daily to Healthy Male and Female Volunteers for 14 Days (27 Doses).

DETAILED DESCRIPTION:
This study is a multiple ascending dose study to Assess the Safety, Tolerability, and Pharmacokinetics of orally dosed PG 760564 Administered Twice Daily to Healthy Male and Female Volunteers for 14 Days (27 Doses). The study is a multiple rising dose (MRD) study of active drug vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and surgically sterile or post-menopausal (last menstrual period > 1 year at the time of enrollment) healthy females, 18-45 years of age, inclusive, at screening;
* Who have not used tobacco or nicotine-containing products within the past 3 months;
* Willing to abstain from caffeine or xanthine-containing beverages, including coffee and tea, chocolate, alcohol, grapefruit juice, and Seville oranges, from 24 hours before admission and for the duration of the study;
* Who have a body mass index (BMI) between 18 and 32 kg/m2.

Exclusion Criteria:

* History of diabetes, cardiovascular, hepatic, renal, or malabsorptive disease;
* History of peptic ulcer disease, hemorrhoids, GI surgery (appendectomy and cholecystectomy are allowed), or GI bleeding;
* History of autoimmune disease;
* History of immunodeficiency or of unusual susceptibility to infectious diseases;
* History of tuberculosis, acquired immunodeficiency syndrome (AIDS), or infection with human immunodeficiency virus (HIV);
* Any history of hypersensitivity or clinically significant allergy to any drug;
* Personal or family history of prolonged QT syndrome or any cardiac conduction abnormality;
* Family history of sudden death;
* History of uveitis or inflammatory ocular disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2005-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S Aronstein, MD, PhD, Study Director — Procter and Gamble
Locations (1):
- Stuart I Harris, MD, PhD, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each Subject enrolled in the study, participated in one period only (e.g., subjects did not start in the 50mg dose group, then proceed to subsequent groups)
Groups:
- Placebo: placebo capsule. This study consisted of 4 sequential periods testing rising doses of PG 760564. Each period randomized participants to receive either placebo or a specific dose of PG 760564. Subjects enrolled in a period participated in that period only.
- 50 mg PG 760564: 50 mg PG 760564 Administered Twice for 14 Days (27 Doses). Subjects enrolled in this period participated in one period only (e.g., subjects did not start in the 50mg dose group, then proceed to subsequent groups)
- 100 mg PG 760564: 100 mg PG 760564 Administered Twice for 14 Days (27 Doses). Subjects enrolled in this period participated in one period only (e.g., subjects did not start in the 100mg dose group, then proceed to subsequent groups)
- 200 mg PG 760564: 200 mg PG 760564 Administered Twice for 14 Days (27 Doses). Subjects enrolled in this period participated in one period only (e.g., subjects did not start in the 200mg dose group, then proceed to subsequent groups)
- 400 mg PG 760564: 400 mg PG 760564 Administered Twice for 14 Days (27 Doses). Subjects enrolled in this period participated in one period only (e.g., subjects did not start in the 400mg dose group, then proceed to subsequent groups)
Period: Period 1 - 50 mg Dose Group
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564
Started | 3 | 8 | 0 | 0 | 0
Completed | 3 | 7 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: Period 2 - 100 mg Dose Group
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564
Started | 3 | 0 | 8 | 0 | 0
Completed | 2 | 0 | 8 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Period: Period 3 - 200 mg Dose Group
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564
Started | 3 | 0 | 0 | 8 | 0
Completed | 3 | 0 | 0 | 8 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4 - 400 mg Dose Group
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564
Started | 4 | 0 | 0 | 0 | 8
Completed | 4 | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564 | Total
Number analyzed (Participants) | 13 | 8 | 8 | 8 | 8 | 45
Age, Categorical [Count of Participants; unit: Participants] — This study consisted of 4 sequential periods testing rising doses of PG 760564. Each period randomized participants to receive either placebo or a specific dose of PG 760564. Subjects enrolled in a single period (i.e., no subject participated in more than one period)
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 13 | 8 | 8 | 8 | 8 | 45
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] — This study consisted of 4 sequential periods testing rising doses of PG 760564. Each period randomized participants to receive either placebo or a specific dose of PG 760564. Subjects enrolled in a single period (i.e., no subject participated in more than one period)
  years | 34.6 (7.3) | 35.0 (5.8) | 29.9 (7.4) | 36.3 (6.5) | 36.9 (5.8) | 34.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants] — This study consisted of 4 sequential periods testing rising doses of PG 760564. Each period randomized participants to receive either placebo or a specific dose of PG 760564. Subjects enrolled in a single period (i.e., no subject participated in more than one period)
  Participants
    Female | 1 | 0 | 0 | 0 | 1 | 2
    Male | 12 | 8 | 8 | 8 | 7 | 43
Region of Enrollment [Number; unit: participants] — This study consisted of 4 sequential periods testing rising doses of PG 760564. Each period randomized participants to receive either placebo or a specific dose of PG 760564. Subjects enrolled in a single period (i.e., no subject participated in more than one period)
  participants
    United States | 13 | 8 | 8 | 8 | 8 | 45

OUTCOME MEASURES:

1. Primary Outcome: AUCτ Over a Dosing Interval (τ = 12 Hours) on Day 14
Description: the area under the plasma concentration-time curve over a dosing interval (τ = 12 hours) on Day 14 of Multiple Dose Oral Administration of PG-760564 Given Every 12 Hours
Time Frame: 14 days
Population: PG 760564 blood plasma concentrations were not measured for the placebo arm
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564
Number analyzed (Participants) | 0 | 7 | 8 | 8 | 4
ng*h/mL |  | 12090.998 (2926.950) | 23472.1329 (9858.248) | 30005.781 (9955.931) | 50354.938 (9781.333)

2. Primary Outcome: Cmax Over a Dosing Interval (τ = 12 Hours)on Day 14
Description: Maximum plasma concentration (Cmax) over a dosing interval (τ = 12 hours)on Day 14
Time Frame: 12 hours on Day 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564
Number analyzed (Participants) | 0 | 7 | 8 | 8 | 4
ng/mL |  | 1601.4 (318.2) | 2951.3 (1148.2) | 3935.0 (953.1) | 7195.0 (279.2)

3. Primary Outcome: Tmax Over a Dosing Interval (τ = 12 Hours) on Day 14
Description: the time at which maximum plasma concentration occurred (Tmax) Over a Dosing Interval (τ = 12 Hours) on Day 14
Time Frame: 12 Hours on Day 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564
Number analyzed (Participants) | 0 | 7 | 8 | 8 | 4
hours |  | 2.46 (0.98) | 2.89 (0.63) | 3.01 (0.54) | 2.03 (0.82)

4. Primary Outcome: t½,z Over a Dosing Interval (τ = 12 Hours)on Day 14
Description: t½,z is the terminal exponential half-life; over a Dosing Interval (τ = 12 Hours)on Day 14
Time Frame: over a Dosing Interval (τ = 12 Hours) on Day 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564
Number analyzed (Participants) | 0 | 7 | 8 | 8 | 4
hours |  | 9.411 (2.640) | 7.882 (1.814) | 10.223 (3.947) | 9.701 (1.714)

ADVERSE EVENTS:
Arm/Group | Placebo | 50 mg PG 760564 | 100 mg PG 760564 | 200 mg PG 760564 | 400 mg PG 760564
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/13 | 7/8 | 7/8 | 8/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | 50 mg PG 760564 (N=8) | 100 mg PG 760564 (N=8) | 200 mg PG 760564 (N=8) | 400 mg PG 760564 (N=8)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Dry (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tenderness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Faecal occult blood positive (Investigations) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6) | 1 (1) | 7 (7) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data, calculations, interpretations, opinions, and recommendations are the property of P&GP. In the event study results are published in the scientific literature by P&GP, acknowledgment will be made to the Investigator(s) in the accepted style, as appropriate.